CLINICAL TRIAL: NCT04026360
Title: Impact of Early Lung Physiology, Viral Infections and the Microbiota on the Development and Progression of Lung Disease in Children With Cystic Fibrosis
Acronym: SCILD
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Children's Hospital, Zurich (Other); Centre Hospitalier Universitaire Vaudois (Other); Kantonsspital Aarau (Other); University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: SCILD
Record Dates: First submitted 2019-05-14; First posted 2019-07-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Confirmed Diagnosis of Cystic Fibrosis
Keywords: Infants; Cystic Fibrosis; Inflammation; Microbiome; Airway growth; Airway development; Genetic predisposition; Tobacco
MeSH Terms: conditions — Cystic Fibrosis; Inflammation; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oropharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
This study collects data on microbiological factors and lung function parameters (e.g. spirometry, body plethysmography, lung-MRI) to assess their interaction on the lung growth and lung development of infants and children with Cystic Fibrosis (CF).

DETAILED DESCRIPTION:
Background:

Cystic fibrosis (CF) is the most common lethal inherited disease in North European populations, affecting approximately 1:2500 live births. It is a multisystem disorder with respiratory morbidity and mortality being the leading cause of death. Lung disease in CF is characterized by neutrophil-dominated inflammation and chronic bacterial infection of the airways, which results in deterioration of lung function and premature death [1]. Despite improved survival in successive birth cohorts, the current median survival age of patients with CF is about 40 years [2]. Understanding the initiating events of CF lung disease (e.g viral infections and microbiome) and their influence on disease progression throughout early childhood is essential to improve survival through targeted early interventions.

Objectives:

The overarching aim of this study is to identify early life predictors of disease progression in children with CF. Therefore, this study implies three objectives, as follows: i) to investigate the effect of respiratory viral infections on microbiota dynamics in the first year of life in infants with CF, and to examine their influence on lung function at 1 year of age; ii) to examine whether deficits in lung function in the first year of life in infants with CF persist to pre- and school age and adolescence and are associated with impaired functional and structural abnormalities at 3, 6, 9, 12, 15 and 18 years of age; and iii) to determine the principal drivers of impaired lung function at 1 year and impaired lung function and structural outcomes at 3, 6, 9, 12, 15 and 18 years of age in individuals with CF.

Methods:

Lung function, magnetic resonance imaging (MRI), respiratory symptoms and quality of life questionnaires, microbiology, medical history and clinical data will be collected during each phase of the study.

Recruitment and participation:

Infants with CF diagnosed by NBS will be recruited at the time of their first lung function test in Bern at the age of 4-8 weeks. As part of the protocol for the diagnosis and follow-up of CF infants diagnosed by NBS, which has been implemented by the Task Force for CF NBS on behalf of the Swiss Working Group for Cystic Fibrosis, optional infant lung function at the University Children's Hospital of Bern is proposed to all parents of newly diagnosed CF infants.

Information collected:

Lung function data:

* Tidal breathing parameters (minute ventilation, respiratory rate, tidal volume, tidal expiratory flow, tidal inspiratory flow, time to peak expiratory flow) averaged over 100 breaths
* Multiple breath washout (FRC, LCI, moment ratios) and single breath washout (molar mass)
* Spirometric forced expiratory volume loops (FVC, FEV1, PEF, MEF50)
* Body plethysmography (airway resistance, lung volumes: TLC, FRC, RV)
* Respiratory Rate over 60 seconds
* Fractional exhaled nitric oxide (marker of airway inflammation)
* Resistance interrupter measurement
* Electric nose
* Forced oscillation technique
* Electrical impedance tomography
* Impedance plethysmography

Microbiological data:

* Nasal swabs (respiratory virus and bacterial diagnostics, as well as host transcriptome analysis)
* Pharyngeal swabs (bacterial colonization and microbiota analysis)
* Sputum (to analyse the neutrophils)

Blood count (hemoglobin concentration, hematocrit, leukocyte number, lymphocyte number, lymphocyte count, eosinophil count, basophil count, monocyte count, promyelocyte count, myelocyte count, platelet count, immunoglobulin E level, interleukins, Granulocyte-Monocyte-Colony Forming Unit, Tumor Necrosis Factor alpha, Interferon gamma and Interferon lambda)

Urine (to estimate the tobacco exposure during pregnancy (amount of Cotinine) and the content of caffeine and steroid profile)

Lung MRI:

Functional and structural images of the lung

Skin-Prick Test (test for pollen, trees, house dust mite, cat and dog)

Questionnaires (to assess quality of life)

Medical history (information on respiratory symptoms, pulmonary exacerbations, hospitalisations and regular therapy)

Study database:

All study data is recorded in an Access-database with SQL Servers by electronic Case Report Forms. The database is accordant to the HFG and was adapted together with the CTU.

Funding:

Schweizerischer Nationalfonds (SNF), Schweizerische Gesellschaft für Cystische Fibrose (CFCH), Departement Lehre und Forschung des Inselspitals Bern

ELIGIBILITY:
Inclusion Criteria:

* Infants with a confirmed diagnosis of CF by NBS
* Age <=18 years
* Written informed consent by patient and/or parent

Exclusion Criteria:

* Need for respiratory support for more than three days
* Severe malformations or known diseases other than CF
* Maternal drug abuse
* Known severe maternal disease
* Severe Problems of communication
* Pacemaker, continuous glucose monitor

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic Fibrosis Patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07-01 (Actual); Primary Completion 2050-08-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Multiple Breath Washout | Every third year from the age of 4-8 weeks/1 year till 18 years.
  Longitudinal assessment of lung volume and ventilation inhomogeneity
Spirometry | Every third year from the age of 4-8 weeks/1 year till 18 years.
  Longitudinal assessment of long volumes.
Body plethysmography | Every third year from the age of 4-8 weeks/1 year till 18 years.
  Longitudinal assessment of ventilation inhomogeneity.
Magnetic Resonance Imaging (MRI) | At the age of 4-8 weeks, 1, 3, 6, 9, 12, 15 and 18 years
  Longitudinal assessment of regional lung perfusion and ventilation
Nasal swabs | At the age of 4-8 weeks, 1, 3, 6, 9, 12, 15 and 18 years
  Longitudinal assessment of viral and bacterial colonization of the nasal swab
Weekly swabs | Weekly from the visit at the age of 4-8 weeks till the age of 1 year
  Respiratory virus and bacterial diagnostic
Swabs during respiratory infection | From the visit at the age of 4-8 weeks till the age of 1 year
  Respiratory viruses and Bacteria, changes of the microbial flora
Routine swabs in CF | At the age of 4-8 weeks, 1 year and at each 3-monthly clinic visit during the age of 3, 6, 9, 12, 15 and 18 years
  Longitudinal assessment of bacterial changes, changes of the resistome (genes conferring antibiotic resistance) and the changes of the microbial flora

SECONDARY OUTCOMES:
Respiratory Rate (RR) | From the visit at the age of 4-8 weeks till the age of 1 year
  The number of breaths over 60 seconds
Sweat test | At the age of 3, 6, 9, 12, 15 and 18 years
  Sweat Chloride concentration

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Latzin, MD PhD, Principal Investigator — University Children's Hospital Bern
Locations (1):
- University Children's Hospital Bern, Bern, Switzerland